CLINICAL TRIAL: NCT05301660
Title: Effect of Nicotine Transdermal Patch on Cognitive Function and Glycolipid Metabolism in Non-smoking Patients With Schizophrenia
Brief Title: Effect of Nicotine Transdermal Patch on Cognitive Function and Glycolipid Metabolism in Non-smoking Schizophrenia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Yanhui Liao, Deputy Chief Physician, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20220111-10
Record Dates: First submitted 2022-02-13; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia
Keywords: nicotine transdermal patch; cognitive function; lycolipid metabolism; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): People with schizophrenic disorders: receiving nicotine transdermal patches.
  Interventions: Drug: Nicotine transdermal patch
- Control group (Placebo Comparator): People with schizophrenic disorders: receive placebo treatment.
  Interventions: Drug: Nicotine transdermal patch

INTERVENTIONS:
Drug: Nicotine transdermal patch — 14 mg / tablet, one tablet a day, attached to the patient's back for 8 weeks
  Other Names: nicotinell

SUMMARY:
Schizophrenia is a group of severe mental disorders of unknown etiology, with significant abnormalities in mental activities such as cognition, thinking, emotion, and behavior, and lead to obvious occupational and social function damage. At present, many studies have found that nicotine and cognitive function changes are related, and many studies have carried out a series of explorations for patients with schizophrenia, but there is no study on the mechanism of nicotine on cognitive function in patients with schizophrenia through changes in glycolipid metabolism, and this study intends to explore whether nicotine participates in the cognitive changes of patients with schizophrenia by regulating glycolipid metabolism, which is conducive to the in-depth study of the mechanism of cognitive function change in schizophrenia, in order to find an effective way to improve the cognitive function of schizophrenia.

DETAILED DESCRIPTION:
The project plans to include 80 non-smoking patients with schizophrenia. If you meet the study enrollment requirements and agree to participate in the study, we will number you and establish a medical record file. During the course of the study, you will be randomly grouped. The intervention group received nicotine transdermal patch (14 mg/tablet) one tablet per day, while the placebo group received a similar-looking placebo patch for a period of 8 weeks. The study was designed to be double-blind, meaning that neither you nor the investigator knew your group until the study was completed. Before and after treatment, you will need to cooperate with the questionnaire assessment, which includes: the subject's general demographic information, medical history, smoking status, nicotine dependence, cognitive function using MCCB (MATRICS Consensus Cognitive Battery) assessment, symptom severity panss (PANSS) assessment, Symptoms of depression and anxiety were assessed using GAD-7 (Generalized Anxiety Disorder) and PHQ-9 (Patient Health Questionnaire-9, PHQ-9).

ELIGIBILITY:
Inclusion Criteria:

1. Using the DSM-V International Neuropsychiatric Jane's Interview Questionnaire (M.I.N.I.);
2. Meet the DSM-V symptom criteria for the diagnosis of schizophrenia;
3. Course of illness for 5 years and less;
4. The cumulative number of cigarettes smoked in the past is less than 100;
5. Lower secondary school or above education level;
6. Han Chinese;
7. years old≥ 18 years old;
8. Right hand;
9. Voluntarily join the study and sign an informed consent form.

Exclusion Criteria:

1. Schizophoratic disorder, bipolar disorder, mental retardation, anxiety spectrum disorder, psychotic disorder caused by drugs, alcohol and other psychoactive substances that meet the diagnostic criteria of DSM-V;
2. Have a history of cerebral organic diseases or head injury;
3. have a history of alcohol and drug dependence;
4. history of impaired consciousness for more than 5 minutes;
5. History of endocrine diseases such as thyroid dysfunction and diabetes mellitus;
6. Those who have serious abnormalities in blood picture, heart, liver and kidney function after examination;
7. pregnant and nursing women;
8. people who have been treated with electroconvulsiveness;
9. There are contraindications to magnetic resonance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-22 (Estimated); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Cognitive function of the subject（score） | 30-40 minutes
  In this study, cognitive function is assessed using the Repeatable Battery for the Assessment of Neuropsychological Status（RBANS）. RBANS measures 5 aspects of neuropsychological function: (1) immediate memory (2) visual spatial structure (3) language (4) attention (5) delayed memory.The higher the score on the assessment scale, the better the cognitive function of the subjects.Scale assessments are done once at baseline and at the end of the 2-week follow-up period, for a total of two tests.
Negative and positive symptoms of the subject（score） | 30-40 minutes
  In this study, negative and positive symptoms in subjects were assessed with Positive and Negative Syndrome Scale（PANSS）.PANSS includes 7 positive scales, 7 negative scales, 16 general psychopathological scales, and 3 supplemental items to assess the risk of attack.The higher the score on the assessment scale, the more severe the subject's symptoms.Scale assessments are done once at baseline and at the end of the 2-week follow-up period, for a total of two tests.
Serum nicotine metabolic rate （%） | 40 minutes
  This study used blood samples from subjects to detect what percentage of nicotine concentrations were available.Subjects were tested once at baseline and after 2 weeks of follow-up, for a total of 2 sessions.
Structural characteristics of the brain (mm) | 30 minutes
  We assessed the brain structure of the subjects by magnetic resonance imaging, once at baseline and once at the end of the 2-week follow-up, for a total of two examinations.We measure how many mm of white matter and gray matter are in the brain.
The function of the subject's brain （mmol/L） | 30 minutes
  We examined the function of the subjects' brains by magnetic resonance imaging, detecting concentrations of metabolites including creatine and creatine phosphate (tCr), glutamate (Glu), inositol (mI), N-acetylbionate (NAA), glycerophosphatecholine (GPC), and glutamic acid and glutamine (Glx).Tests are done at baseline and after 2 weeks of follow-up.
The blood lipid level of the subject（mmol/L） | 1 hour
  The subjects' blood lipid levels included cholesterol, triglycerides, and lipoprotein alpha, in addition to HDL cholesterol and LDL cholesterol.Subjects were tested once at baseline and after 2 weeks of follow-up, for a total of 2 sessions.

SECONDARY OUTCOMES:
The subject's level of depression（score） | 5-10 minutes
  In this study, we used Generalized Anxiety Disorder-7（GAD-7 ）to assess the level of depression in subjects, and the higher the score, the more severe the degree of depression.Scale assessments are done once at baseline and at the end of the 2-week follow-up period, for a total of two tests.
The subject's level of anxiety （score） | 5-10 minutes
  In this study, we used Patient Health Questionnaire-9 （PHQ-9） to assess subjects' anxiety levels, and the higher the score, the more severe the level of anxiety.Scale assessments are done once at baseline and at the end of the 2-week follow-up period, for a total of two tests.
The subject's sleep status （score） | 10-15 minutes
  The study used Pittsburgh sleep quality index（PSQI）to assess the sleep status of the subjects, and the higher the score, the worse the sleep quality.Scale assessments are done once at baseline and at the end of the 2-week follow-up period, for a total of two tests.